CLINICAL TRIAL: NCT05632289
Title: Effects of Osteopathic Treatment in Combination With Usual Care in the Management of Pain Associated With Sickle Cell Disease: A Randomized Controlled Trial.
Brief Title: Osteopathic Manipulation in the Management of Pain Associated With Sickel Cell Disease
Acronym: OSTEODREP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: College Osteopathique de Provence Aix-Marseille (Other)
Collaborators: University Hospital, Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: COPAixMarseille
Record Dates: First submitted 2022-10-28; First posted 2022-11-30 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Sickle Cell Disease
Keywords: osteopathic manipulative treatment; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteopathic treatment (Experimental)
  Interventions: Other: osteopathic manipulative therapy
- sham of osteopathic treatment (Sham Comparator)
  Interventions: Other: sham osteopathic manipulative therapy

INTERVENTIONS:
Other: osteopathic manipulative therapy — osteopathic manipulative therapy : manuel therapy
  Arms: osteopathic treatment
Other: sham osteopathic manipulative therapy — placebo of osteopathic treatment
  Arms: sham of osteopathic treatment

SUMMARY:
Background: Sickle cell disease is the most common monogenic disease in the world caused by a mutation in the β-globin gene which creates abnormal hemoglobin called HbS. This polymer deforms the erythrocyte, making it more fragile and less flexible, thus leading to the occlusion of small blood vessels. This obstruction is the cause of painful vaso-occlusive crises and ischemia-reperfusion phenomena.

Patients with sickle cell disease undergo major acute and chronic pain responsible for a significant deterioration in their quality of life and a significant consumption of analgesics, often daily, sometimes with the development of addictive behavior. Improved analgesic management was associated with improved disease prognosis. Several studies have shown the effectiveness of the osteopathic approach in the management of chronic pain. Our hypothesis is that the association with the standard treatment of osteopathy sessions could improve but also prevent the chronic pain frequent in patients with sickle cell disease.

Objectives: Our main objective is to study the effectiveness of an osteopathic treatment in adult sickle cell patients with chronic pain on the reduction of the consumption of level I and II analgesics at 3 months (D90 +/- 15 days).

Methods/Experimental design: This is a single-blind prospective randomized controlled monocentric study. The study population will be composed of 37 sickle cell patients aged over 18 years. The patients included will be allocated into two groups: one group will receive the osteopathic treatment and the 2nd group will receive the "placebo" treatment. Analgesic consumption will be assessed by weekly self- questionnaire. The evaluation of the pain will be carried out by the visual analogue scale (VAS). The degree of stress will be measured using the Perceived Stress Scale (PSS). Patients will receive an osteopathic treatment or a "placebo" treatment, one session every 4 weeks for 12 weeks with a total of 3 sessions per patient. The duration of each session is 45 minutes. Pain and stress assessments will be done before each session. A final evaluation will be carried out 3 months after the end of the osteopathic or "placebo" treatment. Data analysis will be performed using SPSS version 17.0 software. The significance threshold will be set at 0.05. This is the first protocol that aims to evaluate, with scientific rigor, the impact of the osteopathic approach in the management of pain in patients with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* patients with major sickle cell syndrome
* Suffering from acute or chronic pain
* Aged over 18 and legally responsible
* The informed consent of the patients will be collected

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients who underwent surgery in the 6 months prior to inclusion
* Patients with known medical contraindications to osteopathic manipulations: vertebral compression, severe osteoporosis, progressive osteonecrosis and not treated with a prosthesis
* Patients with acute stroke
* Patients with cerebral arteriovenous malformation or cerebral aneurysm
* Patients participating in another interventional clinical research protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2022-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The consumption of nonopioid and weak opioid analgesics | 3 month
  Analgesic consumption will be assessed by weekly self-questionnaire

SECONDARY OUTCOMES:
pain assessement | 3 month
  Pain assessment will be performed using the Visual Analog Scale score. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Perceived stress assessment | 3 month
  The degree of stress will be measured using the Perceived Stress Scale (PSS). The Perceived Stress Scale (PSS-10) is a 10-item questionnaire originally developed by Cohen et al. (1983) widely used to assess stress levels in young people and adults aged 12 and above. It is a measure of the degree to which situations in one's life are appraised as stressful. Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives.

CONTACTS AND LOCATIONS:
Locations (1):
- Collège Ostéopathique de Provence Aix-Marseille, Marseille, PACA, France

IPD SHARING:
Plan to Share IPD: Undecided